## Patient Identification Number for this trial: Evaluation of the safety and effectiveness of the global treatment including multilayer compression therapy (Urgo KTwo®) in addition to an interactive dressing (UrgoStart® Plus in the management of venous leg ulcers PROTOCOL NUMBER: EUS23-4 IRAS ID: 327680 PROJECT REF NO: 23/003/GHT

Name of Lead Researcher: Mr. Colin Davies, Clinical Lead (Leg Ulcers)

| | | Ple | ease initial<br>box |
|---|---|---|---|
| I confirm that I have read and understand the information sheet dated 25 <sup>th</sup> July 2023 for the above study and have had the opportunity to ask questions. | | | |
| I understand that my participation is volun without giving any reason, without my me | • | • | |
| I understand that relevant sections of my relooked at by Regulatory authorities where I give my permission for these individuals t | it is relevant to my taking part | | |
| I understand that my data will be held on a computer. I give my permission for this data to be held on computer by these parties. | | | |
| I give my permission for you to contact my General Practitioner (GP). | | | |
| I agree to take part in the above study. | | | |
| Name of Patient | Date | Signature | |
| Name of Person taking consent (if different from researcher) | Date | Signature | |
| Mr. Colin DAVIES<br>Researcher | <br>Date | <br>Signature | |

Version 1.4 25<sup>th</sup> July 2023 Page 1/1

<sup>\*1</sup> for patient (copy); 1 for medical notes (copy); 1 for participant's GP (copy); 1 for researcher (original)